CLINICAL TRIAL: NCT03957304
Title: Intranasal Dexmedetomidine for Laceration Repair in Children: a Dose-finding Study
Brief Title: Intranasal Dexmedetomidine Dose-finding Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 51384
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-04

CONDITIONS: Laceration Repair
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Dose-escalation pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of dose levels will not be possible so outcome assessors will be blinded by virtue of being remote from the clinical encounter. Furthermore, video segments will commence immediately after intranasal sprays are given so outcome assessors will not see what volume is administered. Two independent assessors will score each video and an interrater agreement (kappa) will be calculated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexmedetomidine 1 mcg/kg (Experimental): Intranasal dexmedetomidine 100 mcg/mL (Precedex, Pfizer) 1 mcg/kg (max 100 mcg or 1 mL).
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 2 mcg/kg (Active Comparator): Intranasal dexmedetomidine 100 mcg/mL (Precedex, Pfizer) 2 mcg/kg (max 100 mcg or 1 mL).
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 3 mcg/kg (Active Comparator): Intranasal dexmedetomidine 100 mcg/mL (Precedex, Pfizer) 3 mcg/kg (max 100 mcg or 1 mL).
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 4 mcg/kg (Active Comparator): Intranasal dexmedetomidine 100 mcg/mL (Precedex, Pfizer) 4 mcg/kg (max 100 mcg or 1 mL).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal dexmedetomidine

SUMMARY:
The most common injury prompting an emergency department (ED) visit in children is a cut (laceration) that requires repair using stitches or skin glue. Despite anesthetic (freezing), laceration repair is often very distressful because in young children, most occur on the face. There is currently no effective drug to relieve the distress of laceration repair in children. The goal is to find a safe and effective drug to reduce distress in children undergoing laceration repair. Dexmedetomidine is a new drug that safely provides mild sedation and can be given as a painless nasal spray. Intranasal dexmedetomidine (IND) has been shown to reduce distress in children undergoing painful procedures such as dental work and intravenous insertion. However, no large study has explored IND for laceration repair. In order for research to change the way we care for children, a large study that enrolls children across many paediatric EDs needs to be performed. The first step is to conduct a smaller study to identify the safest and most effective dose. The proposed study plans to enroll 55 children age 1-10 years who require laceration repair.

DETAILED DESCRIPTION:
Design: This study will be designed as a phase II single-arm dose-escalation pilot study using the continual reassessment method.

Protocol: Sedation will be measured using the Pediatric Sedation State Scale (PSSS), an instrument validated for video scoring of children undergoing painful procedures. The PSSS is scored from 0 (dangerously sedated) to 5 (least sedated) easily by non-medical personnel and assesses over sedation and under sedation. Adequate sedation is a score of 2 or 3. Participants will be consecutively assigned to increasing doses of IND from 1-4 mcg/kg based on the continual reassessment method. Participants will be assigned to doses of IND from 1-4 mcg/kg, increasing in whole number increments. Initially three participants will receive 1mcg/kg and the number of participants at each dose of IND will be recorded. Data from these participants will be used to update a Bayesian model for the dose-response curve for all three categories of sedation. The following three participants will be assigned the dose with the highest posterior probability of an efficacy close to 0.8. This balances the need to determine the most efficacious dose but prevents an excessive number of over-sedations. For the Bayesian dose response model, a determination will be made as to the overall score category for each participant ("adequate", "over", or "under sedated" based on the PSSS). To be scored as "adequate", a participant must have a PSSS score of 2 or 3 for at least 90% of observations from initial positioning to tying of the last suture. If a participant does not retain a PSSS score of 2 or 3 for at least 90% of the observations, they will be categorized as either over or under-sedated, if the majority of the remaining PSSS scores are 0 or 1 or 4 or 5, respectively. Furthermore, if the participant remains awake, but not distressed during the procedure, they will be scored as a 2 based on the PSSS. However, for the purposes of the Bayesian dose response model, they will be scored as "under sedated" to avoid concluding that a lower dose of IND is effective based on the outcomes for participants that did not require sedation. Finally, participants who are noncompliant with IND will be categorized as an over-sedation as it is assumed that this dose was not well tolerated by the participant and dose escalation should be avoided. Data will be reviewed after each dose increment by a data safety monitoring board, who will confirm it is safe to escalate. Permissible co-interventions include topical and subcutaneous anesthetic, oral or IV analgesics, non-pharmacologic strategies for pain and distress.

Screening and Enrollment: Participants will be consecutively screened for eligibility during the hours of study recruitment.

Sample Size: This was calculated using the Bayesian continual reassessment method (20). Based on an adverse event rate of 10%, 4 dosing levels, an odds ratio for the effect size of 1.8, and a phase II trial accuracy level of 60%, an estimated a sample size of 55 participants was calculated.

ELIGIBILITY:
Inclusion Criteria:

* children age 1-10 years who present to the ED with an isolated laceration < 5 cm
* deemed to require suture repair based on the opinion of the treating physician
* predicted to resist positioning for laceration repair based on the opinion of the caregiver

Exclusion Criteria:

* laceration repair requiring procedural sedation (without IND) or local nerve block, - other injuries requiring reduction (fracture or dislocation) or repair (nailbed injury or laceration)
* lacerations containing foreign body material (including dirt and debris)
* history of hypersensitivity to dexmedetomidine
* occlusion of at least one nare due to mucus, polyps, septal deviation, etc.
* concomitant use of an alpha 2-adrenergic receptor agonist
* bradycardia or hypotension for age (possible transient but clinically insignificant adverse effects of dexmedetomidine)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Adequate sedation | Index visit
  The number of participants with adequate sedation defined as a PSSS or 2 or 3 for the duration of the measurement period (initial positioning to tying of the last suture)

SECONDARY OUTCOMES:
Onset of sedation | Index visit
  Time to adequate sedation (based on PSSS score)
Adverse effects | Index visit
  The number of participants with adverse effects based on the Quebec Guidelines for Reporting of Adverse Effects in Children
Anxiolysis | Index visit
  Degree of anxiolysis as measured using the modified Yale Preoperative Anxiety Scale (mYPAS). The mYPAS is an observationale scale consisting of 22 items across 5 categories. The total score ranges from 0 to 100 with higher scores indicating greater anxiety.
Compliance | Index visit
  Number of participants deemed a compliant with intervention administration
Satisfaction with laceration repair: 5-item Likert scale | Index visit
  Satisfaction score using a 5-item Likert scale obtained from the caregiver, child (if > 7 years), individual performing the repair, and bedside nurse
Nasal irritation | Index visit
  Score on the Faces Pain Scale - Revised (FPS-R) and obtained from children age > 4 years
Length of stay | Index visit
  Duration of time from triage assessment to discharge time
Consent rate | Index visit
  Proportion of eligible participants consented
Delayed maladaptive behaviors | 48 hours post-discharge
  Proportion of children with delayed maladaptive behaviors measured with the Post-Hospital Behavior Questionnaire (PHBQ) assessed 24-48 hours post discharge. The PHBQ is comprised of 27 items among six subscales (general anxiety and regression, separation anxiety, eating disturbance, aggression toward authority, apathy/withdrawal, anxiety about sleep. For each item, parents are asked to compare their child's behavior before hospitalization to their current behavior (post-hospitalization) on a Likert-type scale using the following five response options: much less than before (1), less than before (2), same as before (3), more than before (4), and much more than before (5), producing a range from 27-135 with higher scores indicating greater severity of maladaptive behaviors.
Wound complications | 14 days post-discharge
  Number of participants with wound complications within 14 days of discharge (infection; dehiscence; contracture; retained suture material).

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poonai N, Sabhaney V, Ali S, Stevens H, Bhatt M, Trottier ED, Brahmbhatt S, Coriolano K, Chapman A, Evans N, Mace C, Creene C, Meulendyks S, Heath A. Optimal Dose of Intranasal Dexmedetomidine for Laceration Repair in Children: A Phase II Dose-Ranging Study. Ann Emerg Med. 2023 Aug;82(2):179-190. doi: 10.1016/j.annemergmed.2023.01.023. Epub 2023 Mar 3. PMID 36870890

DOCUMENTS (1):
  • Study Protocol (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03957304/Prot_000.pdf